CLINICAL TRIAL: NCT05653960
Title: The Clinical Outcomes After Endoscopic Mucosal Resection or Endoscopic Submucosal Dissection of Colorectal Neoplasms - A Multicenter Registry
Brief Title: Clinical Outcomes After EMR or ESD of Colorectal Neoplasms - A Multicenter Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2022.474
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenoma
Keywords: Endoscopic mucosal resection; Endoscopic submucosal dissection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — s-formylglutathione hydrolase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who undergo EMR or ESD: Subjects who undergo EMR or ESD for colorectal lesions
  Interventions: Other: EMR or ESD

INTERVENTIONS:
Other: EMR or ESD — Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) are two main endoscopic treatment options for colorectal neoplasms

SUMMARY:
This study aims to establish a multicenter registry platform to capture clinical data from subjects undergoing colorectal EMR and ESD.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common causes of cancer-related death, however its morbidity and mortality can be reduced by colonoscopy screening and endoscopic removal of adenomas or early cancers.[1] Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) are two main endoscopic treatment options for colorectal neoplasms. Despite being a safe and convenient procedure, insufficient resection by EMR can result in a high risk of local recurrence, particularly in lesions ≥ 20 mm. Compared with EMR, ESD facilitates a higher rate of en bloc resection and a lower rate of local recurrence. A recent meta-analysis revealed that the local recurrence rate after colorectal ESD was 1% during a 2-year follow-up period. In addition, ESD can facilitate precise pathological diagnosis to assess the risk of lymph node metastasis of early CRC to judge whether salvage surgery is needed. Although the efficacy of colorectal ESD has been demonstrated, its usage is largely limited by its technical difficulty and risk of complications.

Both short- and long-term data on clinical outcomes and safety profiles for colorectal EMR and ESD are needed. Therefore, this study aims to establish a multicenter registry platform to capture clinical data from subjects undergoing colorectal EMR and ESD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who undergo EMR or ESD for colorectal lesions.

Exclusion Criteria:

* Not applicable.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who undergo EMR or ESD for colorectal lesions.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Curative resection rate of EMR or ESD for colorectal neoplasms | 10 years
  The short- and long-term clinical efficacy outcomes of colorectal EMR or ESD
Adverse event rate of EMR or ESD for colorectal neoplasms | 10 years
  The short- and long-term clinical safety outcomes of colorectal EMR or ESD

CONTACTS AND LOCATIONS:
Overall Officials: Louis Lau, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided